CLINICAL TRIAL: NCT01029418
Title: A Phase 1/2 Study of AZD6244 in Combination With Sorafenib in Advanced Hepatocellular Carcinoma
Brief Title: AZD6244 and Sorafenib in Advanced Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The phase II portion was not conducted due to funding issue.
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Principal Investigator, Choo Su Pin, Senior Consultant, National Cancer Centre, Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-20-HEP
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; hepatocellular carcinoma; liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — AZD 6244; Sorafenib; MEK inhibitor I

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD6244 and sorafenib (Experimental): AZD6244+ sorafenib
  Interventions: Drug: AZD6244 and sorafenib

INTERVENTIONS:
Drug: AZD6244 and sorafenib — dose escalation of AZD6244; sorafenib 400mg bd
  Other Names: AZD6244,; MEK inhibitor,; sorafenib,; Raf kinase inhibitor; nexavar

SUMMARY:
This will be a phase I/II clinical trial testing the combination of sorafenib and AZD6244 in advanced hepatocellular carcinoma with Childs A liver cirrhosis. The aim of the phase I portion is to determine appropriate dose of this drug combination. The phase 2 study will look at effectiveness and safety of this drug combination

DETAILED DESCRIPTION:
Patients with unresectable BCLC Stage B/C hepatocellular carcinoma that is biopsy-proven ( histology or cytology from prior tumor biopsy specimen is acceptable Patients without prior systemic treatment ( chemotherapy or molecular targeted therapy) except prior adjuvant therapy, if given more than 6 months ago Child-Pugh class A only ECOG performance status 0 or 1

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable BCLC Stage B/C hepatocellular carcinoma that is biopsy-proven ( histology or cytology from prior tumor biopsy specimen is acceptable)
* Patients without prior systemic treatment ( chemotherapy or molecular targeted therapy) except prior adjuvant therapy, if given more than 6 months ago
* Patients who had prior local therapy ( TACE; PEI; RFA) more than 4 weeks prior to study entry
* No radiotherapy within 4 weeks before entry
* Child-Pugh class A only ( Appendix A)
* Age 21 years and older
* ECOG performance status 0 or 1 ( Appendix A)
* Life expectancy > 3 months.
* Patients must have normal organ and marrow function as defined below:

Absolute neutrophil count > 1.5 x 109/L;Platelets> 75 x 109/L; Haemoglobin > 9.0g/dl;Total bilirubin < 51umol/L ( 3 mg /dL); AST(SGOT)/ALT(SGPT) < 5 X institutional ULN; Creatinine 1.5 ULN; INR <1.7 or prothrombin time ( PT) <4 seconds above ULN; Left ventricular ejection fraction (LVEF) >50%

* Measurable disease according to RECIST. A lesion which has previously been locally treated (including TACE or RFA) is eligible as long as there is evidence of disease progression
* Suitable for oral administration of drug
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior systemic therapy including sorafenib or a MEK inhibitor or sunitinib or other investigational drugs
* Any prior local therapy ( surgery, radiation therapy, hepatic arterial embolization, or cryoablation) within 4 weeks of study entry.
* Prior liver transplant
* NCI CTCAE grade > 3 hemorrhage within 4 weeks of starting study treatment, or documented variceal hemorrhage of any grade within 12 months of study entry (as documented on endoscopy)
* Presence of esophageal varices (> Grade 2) at risk of bleeding and/or serious or non-healing wound/ulcer ( as documented by endoscopy)
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of study entry
* Patients with underlying inflammatory bowel disease, partial or complete bowel obstruction or chronic diarrhea
* Any of the following within the 12 months prior to study drug administration: severe/unstable angina, myocardial infarction, coronary artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, including transient ischemic attack, or pulmonary embolism.
* History of cardiac disease:
* active congestive heart failure
* cardiac arrythmias of NCI CTCAE grade >2 or requiring pacemaker
* uncontrolled hypertension
* cardiomyopathy
* atrial fibrillation rate >100bpm
* Patients with factors that increase the risk of QT prolongation or arrhythmic events ( hypokalemia, family history of long QT interval syndrome) or QTc interval of > 450ms for males or > 470ms for females on screening

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-11; Primary Completion 2014-02 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLT) of the combination of AZD6244 and sorafenib in patients with advanced hepatocellular cancer. | 12-15months

SECONDARY OUTCOMES:
To investigate if the combination sorafenib and AZD6244 increases Time To Progression (TTP) over sorafenib alone in patients with advanced hepatocellular carcinoma patients. | 2-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Su Pin Choo, Principal Investigator — National Cancer Centre, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital Singapore, Singapore
  - National Cancer Centre Singapore, Singapore

REFERENCES:
- [Background] Huynh H, Ngo VC, Koong HN, Poon D, Choo SP, Toh HC, Thng CH, Chow P, Ong HS, Chung A, Goh BC, Smith PD, Soo KC. AZD6244 enhances the anti-tumor activity of sorafenib in ectopic and orthotopic models of human hepatocellular carcinoma (HCC). J Hepatol. 2010 Jan;52(1):79-87. doi: 10.1016/j.jhep.2009.10.008. Epub 2009 Oct 28. PMID 19910069
- [Derived] Tai WM, Yong WP, Lim C, Low LS, Tham CK, Koh TS, Ng QS, Wang WW, Wang LZ, Hartano S, Thng CH, Huynh H, Lim KT, Toh HC, Goh BC, Choo SP. A phase Ib study of selumetinib (AZD6244, ARRY-142886) in combination with sorafenib in advanced hepatocellular carcinoma (HCC). Ann Oncol. 2016 Dec;27(12):2210-2215. doi: 10.1093/annonc/mdw415. Epub 2016 Sep 28. PMID 27681866